CLINICAL TRIAL: NCT01103817
Title: Influence of Vitamin D on Vascular Function in Adolescents and Young Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Farid Mahmud, Staff Physician, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000014567
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes; Adolescents and Young Adults; Vitamin D; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Cardiovascular Diseases | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D Sufficient (No Intervention): Sufficient is defined as a 25 OH vitamin D level >50 nmol/l measured at baseline. No clinical intervention will be assigned to this group.
  Subjects will have fasting bloodwork done. Other study measurements to be taken include: height and weight, stage of puberty, blood pressure, vitamin D and calcium intake information, diabetes risk information, demographic information and spot urine sample.
  We will also do a non-invasive test called a "PAT" or 'peripheral arterial tonometry' to look at the health of your blood vessels.
- Vitamin D Deficient (Experimental): Deficient is defined as a 25 OH vitamin D level ≤ 37.5 nmol/l. This group will receive Vitamin D.
  Subjects will have fasting bloodwork done. Other study measurements to be taken include: height and weight, stage of puberty, blood pressure, vitamin D and calcium intake information, diabetes risk information, demographic information and spot urine sample.
  We will also do a non-invasive test called a "PAT" or 'peripheral arterial tonometry' to look at the health of your blood vessels.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Dosing If the 25 OH Vitamin D level at Baseline/Screening is less than 20 nmol/L then the subject will receive 2000 IU daily.
  If the 25 OH Vitamin D level at Baseline/Screening is between 20 and 37.5 nmol/L then the subject will receive 1000 IU daily.
  Other Names: Ddrops®
  Arms: Vitamin D Deficient

SUMMARY:
The purpose of this study is to study the role of low vitamin D levels on the health of blood vessels or vascular function in adolescents and young adults with type 1 diabetes.

DETAILED DESCRIPTION:
Vitamin D deficiency is known to be common in patients with type 1 diabetes. Studies in adults have shown that vitamin D deficiency is associated with cardiovascular events such as stroke, myocardial infarction and peripheral arterial disease. However, the impact of this deficiency on vascular health in adolescents with diabetes has not been examined. Furthermore given that endothelial dysfunction is reversible, early detection of this process may have therapeutic and prognostic implications in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 1 diabetes, according to Canadian Diabetes Association guidelines
2. Diagnosed with type 1 diabetes for at least 2 years
3. Between the ages of 12 and 18 years

Exclusion Criteria:

1. Previous organ transplantation
2. Diagnosed with familial hypercholesterolemia
3. Active smoker
4. Receiving lipid lowering medications
5. Receiving anti hypertensive medication
6. Significant chronic medical illness, including granulomatous disease
7. History of hypertension
8. BMI >95%tile
9. Known renal failure
10. HbA1c greater than 12% on two successive occasions
11. Known peripheral vascular disease
12. Known hypercalcemia

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Endothelial Function | Baseline
  We will compare endothelial function in adolescents with type 1 diabetes divided into 2 groups on the basis of vitamin D status (deficient and sufficient).
  Endothelial function will be assessed by peripheral arterial tonometry (PAT) which measures the elasticity of the arteries.
Change in Endothelial Function after Treatment with Vitamin D | Baseline, 3 or 6 months
  We will measure the change in endothelial function from baseline in the children that were vitamin D deficient. This measurement will be done once the child has become vitamin D sufficient.
  Vitamin D status will be assessed at 3 months. If the levels remain deficient treatment would continue for another 3 months, with repeat testing at 6 months.
  Endothelial function will be assessed by peripheral arterial tonometry (PAT) which measures the elasticity of the arteries.

SECONDARY OUTCOMES:
Monitoring of Vitamin D Levels in Vitamin D deficient subjects | 2-3 months
  At a vist to take place at 2-3 months, the Vitamin D deficient sujects will undergo blood sampling for 25 hydroxyvitamin D levels to ensure appropriate treatment with D Drops to normalize 25 OH vitamin D levels greater than 50 nmol/L.
Monitoring of Calcium Creatine Ratio in Vitamin D deficient subjects | 2-3 months
  At a vist to take place at 2-3 months, the Vitamin D deficient sujects will have a urine assessment of spot calcium creatinine ratio to ensure that hypercalcemia (calcium/ creatinine ratio greater than 0.7) is not present.
Comparison of Systemic Blood Pressure | Baseline
  We will compare endothelial function in adolescents with type 1 diabetes divided into 2 groups on the basis of vitamin D status (deficient and sufficient).
Comparison of Urinary Albumin/Creatinine Ratio | Baseline
  We will compare the urinary albumin/creatinine ratio in adolescents with type 1 diabetes divided into 2 groups on the basis of vitamin D status (deficient and sufficient).

CONTACTS AND LOCATIONS:
Overall Officials: Farid Mahmud, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada